CLINICAL TRIAL: NCT03791658
Title: Assessment of Adherence to Controller Inhalation Medication in Asthma- and COPD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Lisa Nicky Vancampenhout, Medical student, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PNE 2018-386
Record Dates: First submitted 2018-12-31; First posted 2019-01-02 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Asthma; COPD; Adherence, Medication
Keywords: TAI; Test for the Adherence to Inhalers
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Cross-sectional, single center, single visit study.
  1 group of 70 asthmatics, 1 group of 70 COPD-patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthmatics (Other): From the patients file the following information will be collected by the investigators:
  * Age
  * Sex
  * FEV1 derived from the last spirometry (including spirometry performed on day of study visit).
  * GINA step (Global Initiative for Asthma).
  * Number of exacerbations in the year prior to the study.
  * The prescribed medication: type of inhaler, number of inhalers for maintenance treatment, number of inhalations a day.
  * Number of different medications taken by the patient on a daily basis, excluding the inhalers for maintenance treatment of asthma.
  * FENO (Fraction Exhaled Nitric Oxide) from the day of the study visit (if available).
  Patients will fill out:
  * The 12-question TAI-questionnaire (test for the adherence to inhalers)
  * The Asthma Control Test (ACT)
  Interventions: Other: The 12-question TAI; Other: Information from patients file; Other: The Asthma Control Test (ACT)
- COPD-patients (Other): From the patients file the following information will be collected by the investigators:
  * Age
  * Sex
  * Pack Years
  * GOLD stage (Global Initiative for Chronic Obstructive Lung Disease)(post-bronchodilator FEV1)
  * Number of exacerbations in the year prior to the study.
  * The prescribed medication: type of inhaler, number of inhalers for maintenance treatment, number of inhalations a day.
  * Number of different medications taken by the patient on a daily basis, excluding the inhalers for maintenance treatment of COPD.
  Patients will fill out:
  * The 12-question TAI-questionnaire (test for the adherence to inhalers)
  * The COPD Assessment Test (CAT)
  Interventions: Other: The 12-question TAI; Other: Information from patients file; Other: The COPD Assessment Test (CAT)

INTERVENTIONS:
Other: The 12-question TAI — The 12-question TAI (Test for the Adherence to Inhalers) yields a score indicating level of adherence (high, intermediate or poor). The TAI also provides some indication about the possible mechanisms of non-adherence (sporadic, deliberate or unconscious).
Other: Information from patients file — Depending on which arm or group specific information will be gathered from the patients file after informed consent.
Other: The Asthma Control Test (ACT) — An international validated questionnaire on the symptoms an asthmatic experiences and the disease control in the patient. Only for the Asthmatics arm of the study
  Arms: Asthmatics
Other: The COPD Assessment Test (CAT) — An international validated questionnaire on the symptoms a COPD-patient experiences and the disease control in the patient. Only for the COPD arm of the study
  Arms: COPD-patients

SUMMARY:
The main aim of the study is to evaluate the adherence to controller inhalation medication in asthma and Chronic Obstructive Pulmonary Disease (COPD) in Universitair Ziekenhuis Brussel. Adherence will be assessed using the 12-question Test for the Adherence to Inhalers (TAI) yielding a score indicating level of adherence (high, intermediate or poor). The TAI also provides some indication about the possible mechanisms of non-adherence (sporadic, deliberate or unconscious). The aim of the study is also to compare the adherence between the 2 study subgroups (asthma and COPD patients). Several other factors which could influence the compliance of the patients will also be evaluated: age, sex, pack years, FEV1 (Forced Expiratory Volume 1), exacerbation history, symptom control, type of inhaler and number of inhalers. By identifying different patient and treatment characteristics that lead to non-adherence, future education efforts could be better targeted to these patients presenting the most important unmet need in terms of adherence.

DETAILED DESCRIPTION:
Adherence to the controller inhalation medication is an important component of asthma and COPD care. Good adherence to the prescribed medication is asthma patients is associated with better symptom control and improved lung function. Also, lower exacerbation rate and mortality risk, less healthcare utilisation, lower healthcare-associated costs and a better quality of life are linked with better adherence in asthma and COPD patients.

However, studies have shown that the adherence to therapy in chronically ill patients averages around 50%. In asthma patients the level of adherence varies between 30-70%, while compliance rate in COPD patients is around 20-60% (though the numbers vary). Adherence in asthma and COPD patients is thus generally low.

Adherence in these patients is measured in studies in different ways: electronic device monitoring, dispensing data, drug levels or several self-administered questionnaires, among others. Each technique has its own benefits and drawbacks. However, the easiest to use are the self-administered questionnaires. Although many of these exist, a particularly interesting questionnaire is the TAI (Test for the Adherence to Inhalers). It exists in 2 versions: a 10-question and a longer 12-question test. The 12 question TAI has 2 added questions, in which a healthcare professional evaluates the use of the inhaler by the patient. All 12 questions can then be used to identify different non-compliance behavioural patterns. The advantages of this questionnaire are therefore that it can be used for both asthma and COPD patients, that it is designed specifically for inhalation medication and that it not only measures adherence but also the type of non-compliance .

The main aim of the study is thus to evaluate the adherence to controller inhalation medication in asthma and COPD in Universitair Ziekenhuis Brussel. Adherence will be assessed using the 12-question TAI (Test for the Adherence to Inhalers). The aim of the study is also to compare the adherence between the 2 study subgroups (asthma and COPD patients). Several other factors which could influence the compliance of the patients will also be evaluated: age, sex, pack years, FEV1, exacerbation history, symptom control, type of inhaler and number of inhalers. By identifying different patient and treatment characteristics that lead to non-adherence, future education efforts could be better targeted to these patients presenting the most important unmet need in terms of adherence.

Patient recruitment will take place at the Universitair Ziekenhuis Brussel respiratory outpatient clinic. Before their scheduled appointment, patients they will be screened to participate in the study. Recruitment will start January 2019 until March 2019, or until the target number of patients is reached. On the day of their appointment, the participants will receive all necessary information about the study and the informed consent process from the principal investigator.

Patients will have sufficient time to reflect on their participation in this study and to ask questions. After obtaining the written informed consent from the patients, the necessary interventions (filling in questionnaires and gathering information from the patients files) will take place.

It will be allowed for the patients to provide informed consent and to participate in the study on a later date.

Statistical analysis:

The statistical analysis will be conducted in 3 steps :

1. Preliminary one-way ANOVA to evaluate the dependent variable (TAI level of adherence) for each independent variable.
2. A multi-way ANOVA model will be constructed to include the relevant independent variables and potential two-way interactions, by maximization of adjusted R2 obtained through a backward elimination in order to correct for multicollinearity.
3. In a final step, the model residuals will be checked to satisfy the normality condition through application of the Kolmogorov-Smirnov and Shapiro-Wilk tests, also exploring the influence of potential heteroscedasticity.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatics with treatment ≥ GINA step 2.
* COPD-patients , GOLD stage II-IV.

Exclusion Criteria:

* No spirometry results available.
* COPD patients not on long-acting bronchodilators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Adherence to inhalation medication evaluated using the Test for the Adherence to Inhalers | 15 minutes
  Level of adherence: high (=50 points), intermediate (between 46 and 49 points) or poor (< or = 45 points) .

SECONDARY OUTCOMES:
Type of non-adherence/ Behavioural pattern (using TAI) | 15 minutes
  Sporadic non-adherence: items 1 to 5 <25points Deliberate non-adherence: items 6 to 10 < 25 points Unconscious non-adherence: items 11 and 12 < 4 points
Adherence in correlation to specific factors | 15 minutes
  Asthma patients: Age, sex, FEV1 derived from the last spirometry (including spirometry performed on day of study visit), GINA step, number of exacerbations in the year prior to the study, the prescribed medication: type of inhaler, number of inhalers for maintenance treatment, number of inhalations a day, number of different medications taken by the patient on a daily basis (excluding the inhalers for maintenance treatment of asthma), FENO from the day of the study visit (if available), result of ACT. COPD-patients: Age, sex, Pack Years, GOLD stage and GOLD group, the prescribed medication: type of inhaler, number of inhalers for maintenance treatment, number of inhalations a day, number of different medications taken by the patient on a daily basis (excluding the inhalers for maintenance treatment of COPD).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa N Vancampenhout, Principal Investigator — Master student in Medicine at Vrije Universiteit Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
Choice made with regards to the current General Data Protection Regulation in Europe.

REFERENCES:
- [Background] Plaza V, Fernandez-Rodriguez C, Melero C, Cosio BG, Entrenas LM, de Llano LP, Gutierrez-Pereyra F, Tarragona E, Palomino R, Lopez-Vina A; TAI Study Group. Validation of the 'Test of the Adherence to Inhalers' (TAI) for Asthma and COPD Patients. J Aerosol Med Pulm Drug Deliv. 2016 Apr;29(2):142-52. doi: 10.1089/jamp.2015.1212. Epub 2015 Jul 31. PMID 26230150
- See also: The Asthma Control Test used in this study — http://www.asthmacontroltest.com/
- See also: The COPD Assessment Test used in this study — http://www.catestonline.org/